CLINICAL TRIAL: NCT05316389
Title: Minimal Harvest Dorsalis Major Flap Breast Reconstruction: Retrospective and Prospective Evaluation of Scapulohumeral Comfort, Aesthetic Result and Quality of Life
Brief Title: Retrospective and Prospective Evaluation of Scapulohumeral Comfort, Aesthetic Result and Quality of Life
Acronym: QUARLAMI
Status: Recruiting | Type: Observational
Sponsor: Institut Cancerologie de l'Ouest (Other)
Responsible Party: Sponsor
Other Study IDs: ICO-2021-05
Record Dates: First submitted 2022-03-11; First posted 2022-04-07 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Mammaplasty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- A Retrospective: A = retrospective cohort including all patients treated at the ICO Angers between January 2017 and September 2021
  Interventions: Procedure: Breast reconstruction
- B Prospective: B = prospective including all patients treated at the ICO from February 2022 (2 years of recruitment)
  Interventions: Procedure: Breast reconstruction

INTERVENTIONS:
Procedure: Breast reconstruction — Muscle sparing Latissimus Dorsi Flap or prothesis

SUMMARY:
The dorsalis major flap is an interesting therapeutic option in breast reconstruction because of reliability and reproducibility.

In recent years, the minimal flap technique has been developed, which consists of removing only a portion of the of the large dorsal muscle to reduce the painful and functional sequelae of this surgery.

The objective of this prospective study is to evaluate the functional and aesthetic results in patients who have undergone who have undergone this procedure (prospective cohort) or who will undergo this procedure or prosthetic reconstruction (prospective cohort).

The investigators also wish to evaluate the quality of life of patients after reconstruction with a minimal harvest dorsalis flap or a prosthesis or prosthesis in the prospective cohort.

DETAILED DESCRIPTION:
Retrospective Cohort :

* Clinical data reconstruction and follow-up up to 1 year
* DASH questionnaire
* Breast Q
* aesthetic evaluation (patient and surgeon and other health professional)

Prospective Cohort :

* Clinical data reconstruction and follow-up up to 1 year
* DASH questionnaire (pre-op, at 6 month and at 12 month)
* Breast Q(pre-op, at 6 month and at 12 month)
* aesthetic evaluation (patient and surgeon and other health professional) (at 6 month and at 12 month)

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a desire for breast reconstruction
2. Indication for mastectomy or with a history of mastectomy, with or without preservation of the skin skin,
3. Breast reconstruction procedure by LDPM performed between January 2017 and September2021, (retrospective cohort )
4. Breast reconstruction procedure by LDPM or by prosthesis performed from February 2022 (prospective cohort)
5. Information to the patient and collection of her non-opposition
6. Affiliation to a social security system, or beneficiary of such a system

Exclusion Criteria:

1. Performance of a breast reconstruction by a technique other than LDPM or prosthesis
2. Patient opposed to the use of her data for research
3. Person in an emergency situation, adult subject to a legal protection measure (adult under guardianship, curatorship or safeguard of justice), or unable to express his consent,
4. Impossibility to submit to the medical follow-up of the trial for geographical, social or psychological psychological reasons.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients at the ICO Angers site with an indication for immediate or deferred breast reconstruction for their breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-02-21 (Actual); Primary Completion 2025-02-21 (Estimated); Study Completion 2025-02-21 (Estimated)

PRIMARY OUTCOMES:
functional evaluation of the shoulder and upper limb (mobility and pain) | 6 month
  Disabilities of the Arm, Shoulder and Hand (DASH) (0 = no disability to 100 = maximum disability)

SECONDARY OUTCOMES:
satisfaction of aesthetic by the patient and by the surgeon | 6 month
  5 numerical scales (from 0 to 5) measuring overall satisfaction with the reconstruction, general appearance of the breast, breast shape, breast consistency and breast volume
occurrence of postoperative complications | 6 month
  complications
quality of life through the Breast-Q questionnaire | 6 months
  Breast-Q questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Julia DE FREITAS, Principal Investigator — ICO
Locations (1):
- Institut de Cancerologie de L'Ouest (Ico), Angers, France

IPD SHARING:
Plan to Share IPD: No